CLINICAL TRIAL: NCT03507192
Title: Effects of Muscle Relaxation on Cognitive Function in Patients With Mild Cognitive Impairment and Early Stage Dementia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-05-135
Record Dates: First submitted 2018-04-15; First posted 2018-04-24 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Dementia
Keywords: MCI, Alzheimer's disease, muscle relaxation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (No Intervention): 30 subjects In arm 1, no intervention is performed.
- Arm 2 (Active Comparator): 30 patients In arm 2 , active comparators, Muscle relaxation using full body massage machine is performed every morning and evening for 30 minutes.
  Interventions: Device: Muscle relaxation using full body massage machine

INTERVENTIONS:
Device: Muscle relaxation using full body massage machine — Receiving muscle relaxation machine massage every morning and evening for 30 minutes during a year
  Arms: Arm 2

SUMMARY:
Muscle relaxation has been reported to be effective in alleviating anxiety and agitation symptoms in patients with dementia, but no studies have examined the effects of muscle relaxation therapy on cognitive function changes.

Therefore, the purpose of this study is to compare and validate the improvement of cognitive function in patients with mild cognitive impairment and early alzheimer's dementia aged 50 to 85 years after performing muscle relaxation machine massage regularly.

DETAILED DESCRIPTION:
The prevalence of dementia is approximately 5-10% in the elderly who are over 65 years of age. In Korea, the prevalence of dementia among elderly people aged 65 and over was 9.18% in 2012, and the number of patients with dementia was estimated to be 540,755 (155,955 for male, 384,800 for female). The number of patients with dementia will be doubled every 20 years until 2050, which is estimated to be 840,000 in 2020, about 1.27 million in 2030, and 2.71 million in 2050. Alzheimer's disease is the most common cause of dementia, accounting for 55-70% of all dementia. Major risk factors include age, genetic factors, apolipoprotein E gene, female and brain trauma, but stress is also associated with increased risk of Alzheimer's disease.

Stress can be present anywhere in our daily lives, and stress can energize life, but if people are exposed to stress for a long time, they may develop physical symptoms. Severe and long-term stress can cause or exacerbate diseases such as angina, stroke, hypertension, diabetes, tension headache, back pain, irritable bowel syndrome, asthma and arthritis. Studies about the relationship between stress and Alzheimer's disease have shown that the corticotrophin releasing factor secreted when exposed to stress can increase brain toxic protein such as beta amyloid plaques that are known to be responsible for dementia.

There are various ways to overcome stress, like meditation, yoga and relaxation training methods that individuals can do at home. Relaxation training methods include relaxation using breathing and progressive muscle relaxation. Progressive muscle relaxation therapy stabilizes anxious psychology by stretching and relaxing several muscles of the body in turn. Muscle relaxation promotes arterial and venous flow, lymphatic flow, reduces edema of muscles and connective tissues, and improves organ function to aid homeostasis.

Muscle relaxation has been reported to be effective in alleviating anxiety and agitation symptoms in patients with dementia, but no studies have examined the effects of muscle relaxation therapy on cognitive function changes.

Therefore, the purpose of this study is to compare and validate the improvement of cognitive function in patients with mild cognitive impairment and early alzheimer's dementia aged 50 to 85 years after performing muscle relaxation machine massage regularly.

ELIGIBILITY:
1. Inclusion Criteria (1) Subjects aged 50 to 85 years who understand and agree to the purpose of the study (2) mild cognitive impairment or early stage of Alzheimer dementia (3) CDR of 0.5~1
2. Exclusion Criteria (1) severe cerebral white matter hyperintensities on brain MRI : defined as deep white matter ≥ 2.5 cm, caps or band ≥ 1.0 cm (2) cancer or severe medical illness (3) fear of magnetic resonance imaging (MRI) examination (claustrophobia) (4) MRI contrast agent side effects (4) pacemaker or a metal material which can not be detached (prosthetics, braces, etc.)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
cortical thickiness in 3D MRI | One year after receiving muscle relaxation massage everyday.
  changes of cerebral cortical thickness in 3D MRI

SECONDARY OUTCOMES:
functional connectivity in functional MRI | One year after receiving muscle relaxation massage everyday.
  functional connectivity of default mode network in and resting state fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Sang Won Seo, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Neurology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim YJ, Kim HR, Jung YH, Park YH, Seo SW. Effects of Electrical Automatic Massage on Cognition and Sleep Quality in Alzheimer's Disease Spectrum Patients: A Randomized Controlled Trial. Yonsei Med J. 2021 Aug;62(8):717-725. doi: 10.3349/ymj.2021.62.8.717. PMID 34296549